CLINICAL TRIAL: NCT06032806
Title: Effects of 8 Weeks Moderate and High Intensity Training on Hemoglobin Levels of Female Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Tanzeela Rehman 41008
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Moderate and High Intensity Training and Hemoglobin Levels
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Moderate Intensity) (Experimental): Warm up protocol to reach max HR 50% than moderate intensity exercise. Group A will be given moderate intensity exercise i.e Brisk walk (HR will be in between 50-60% of max HR) .
  Interventions: Other: moderate intensity
- Group B (High Intensity) (Experimental): Warm up protocol achieve 70% of max HR. Group B will be given high intensity exercise i.e Skipping rope (HR will be in between 70-85% of max HR).
  Interventions: Other: High intensity

INTERVENTIONS:
Other: moderate intensity — * Arm circles
  * Leg swings
  * Lunges
  Arms: Group A (Moderate Intensity)
Other: High intensity — * Arm circles
  * Leg swings
  * Lunges
  * Butt kicks
  Arms: Group B (High Intensity)

SUMMARY:
This study aimed to assess the effectiveness of 8 weeks of moderate and high intensity training on hemoglobin levels of female students

DETAILED DESCRIPTION:
Anemia is a global health problem and occurs at all stages of the life cycle but is more prevalent among 50% young females of reproductive age and 21% of age group 9-29 years, faces the same problem in Punjab, a province of Pakistan. Higher percentage was found in hostilities (39.2%) as compared to day scholars (23.1%). Anemia has been shown affect to mental development and learning capacity, stress level, may cause irritability, fatigue, difficulty with concentration, lethargy, weakness, and increased susceptibility to infection. Consequently, anemic patients may tend to be poor in quality of life.

Adult men and adult women have different hemoglobin levels in health. This difference is independent of iron status - iron replete pre-menopausal women have mean hemoglobin levels approximately 12% lower than age & race matched men. National Health and Nutrition Examination Survey (NHANES HI) showed that 9% to11% of adolescent girls and women of child-bearing age were iron-deficient and 2% to5% of them were diagnosed with iron deficiency anemia. Iron deficiency with the presence of low hemoglobin is the criterion for the diagnosis of iron deficiency anemia.There have been frequent reports of a sub-optimal hematological status being observed in athletes involved in intensive physical activity.

Physical activity especially moderate and high intensity reduce mortality and prevent many chronic diseases such as hypertension, diabetes, stroke, and cancer, and stimulate erythropoiesis, which can promote healthy cognitive and psycho-social function and increased hemoglobin concentration Hb lead to increase maximum oxygen carrying capacity. A study reported that aerobic exercise increased hemoglobin (Hb) concentration and hematologic factors in young females.

Recently, the rising prevalence of physical inactivity worldwide has become a major public health concern, and more than one in four adults fail to follow the minimum recommended levels of participating in 150 min of moderate physical activity (MPA) per week.

This is because the network or cell will need more oxygen when doing activities so that there is adaptation in binding oxygen in the blood. But another study conducted on sedentary women suggest that exercise reduce the red blood cells (RBC), hemoglobin (Hb), and hematocrit (Hct) in sedentary women.

Recently, the prevalence and popularity of high intensity interval exercise (HIIE) among young adults has provided an exciting type of exercise and health promotion intervention. High-intensity interval training (HIT) consisting of short bouts of vigorous intensity exercise, interspersed with low-intensity recovery periods, seems to be the most effective method to improve exercise performance not only in well-trained athletes but also in sedentary and diseased individuals.

Literature shows that there isn't any defined physical activity, which can affect the Hb concentration. Currently no study was found in Pakistan regarding effectiveness of Physical activity on Hemoglobin concentration in young female. Internationally there is also conflicting result about the effect of exercise in increasing or decreasing Hb level. The authors conclude that both high and moderate intensity exercises can improve HB levels in female students. They suggest that the benefits of exercise on HB concentration appear to be more pronounced in those with lower baseline HB levels.

Most of the literature showed that level of physical activity is associated with Hb level. But there is paucity in the literature regarding the cause-and-effect relationship of PA and Hb and any defined physical activity, which can affect the Hb concentration in young female. So objective of the current study is to determine and compare the effectiveness of moderate and vigorous physical activity improving hemoglobin concentration in young female.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-25 years.
* Hb levels greater than 10 & less than 12.0 gm/dl

Exclusion Criteria:

* Female staff of the institute.
* Students already engaged in physical activity.
* Hb levels greater than 12.0 & less than 10 gm/dl
* Female having any bony deformity (spine, hip, knee & ankle)

Ages: 23 Years to 27 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
hemoglobin (Hb) level improvement | 8 weeks
  Changes from the baseline will be measured The amount of hemoglobin in whole blood is expressed in grams per deciliter (g/dl). The normal Hb level for males is 14 to 18 g/dl; that for females is 12 to 16 g/dl.
CBC (Complete blood count) | 8 weeks
  Changes from the baseline will be measured The CBC test identifies and counts the 7 types of cells found in the blood, red blood cell, neutrophil, eosinophil, basophil, lymphocyte, monocyte, and platelet.
Pulse oximeter for Heart Rate | 8 weeks
  Pulse oximeters are often used for estimating heart rate at rest and during exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Tanzeela Rehman, DPT, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Sargodha institute of health sciences, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No